CLINICAL TRIAL: NCT01247051
Title: Comparison of Two Different Heart-lung Machine Filling Methods: Precoating Versus Colloidal Fluids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Arndt-H. Kiessling, Head cardiovascular research, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRE001AHK
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Priming; Cardiac Surgery; Cardio Pulmonary Bypass
Keywords: priming; cardiac surgery; cardio pulmonary bypass; precoating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Precoating (Experimental)
  Interventions: Procedure: Precoating
- Standard priming (Active Comparator)
  Interventions: Procedure: Standard priming

INTERVENTIONS:
Procedure: Precoating — preoperative filling of heart lung machine with patients blood
  Arms: Precoating
Procedure: Standard priming — preoperative filling of heart lung machine with colloids
  Arms: Standard priming

SUMMARY:
The study is a single-center, randomized, un-blinded treatment study in which patients (>78 years) with the use off a heart-lung machine were provided into two study arms.

Patient wit "precoating" have a filling of the machine with their own blood. In the comparator arm, a standard priming is used.

ELIGIBILITY:
Inclusion Criteria:

* Age > 78 years
* CPB

Exclusion Criteria:

* Hb <12 mg/dl
* Off pump surgery

Ages: 78 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
blood loss | 24 hours

SECONDARY OUTCOMES:
Inflammatory response | one week

CONTACTS AND LOCATIONS:
Locations (1):
- Goethe University, Frankfurt am Main, Hesse, Germany